CLINICAL TRIAL: NCT02776605
Title: Concurrent Ponatinib With Chemotherapy for Young Adults With Newly Diagnosed Philadelphia Chromosome Positive Acute Lymphoblastic Leukemia
Brief Title: Ponatinib With Chemotherapy for Young Adults Ph Positive Acute Lymphoblastic Leukemia
Acronym: PONALFIL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: PETHEMA Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PONALFIL
Record Dates: First submitted 2016-05-16; First posted 2016-05-18 (Estimated); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: ALL
MeSH Terms: interventions — Prednisone; Vincristine; Daunorubicin; ponatinib; Mercaptopurine; Methotrexate; Etoposide; Cytarabine; Transplantation, Autologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ponatinib (Experimental): 1. Pre-phase (maximum 7 days, -7 to -1) with Prednisone and triple intrathecal therapy (TIT)
  2. Induction (day 1 to day 28 or up to hematological recovery) Vincristine (VCR): 1.5 mg/m2 IV days 1, 8, 15 and 22. Daunorubicin (DNR): 45 mg/m2 IV days 1, 8, 15 and 22. Prednisone (PDN): 60 mg/m2/day, IV or PO, days 1 to 27. Ponatinib 30 mg, PO from day 1 to consolidation. TIT, days 1 and 22.
  3. Consolidation Mercaptopurine (MP): 50 mg/m2, PO days 1 to 7, 28 to 35 and 56 to 63. MTX: 1,5 g/m2, IV days 1, 28 and 56. VP-16: 100 mg/m2/12 h, IV, days 14 and 42. ARA-C: 1000 mg/m2/12 h, IV, days 14-15 and 42-43. TIT days 1, 28 and 56. Ponatinib 30 mg/d PO, from day 1 to day 7 before HSCT".
  4. HSCT (performed ideally within 1 month from the end of consolidation).
  5. Post HSCT therapy (MRD monitoring)
  Interventions: Drug: Prednisone; Drug: Vincristine; Drug: Daunorubicin; Drug: Ponatinib; Drug: Mercaptopurine; Drug: Methotrexate; Drug: VP-16; Drug: ARA-C:; Drug: TIT; Procedure: Autologous transplantation; Procedure: Allo transplantation

INTERVENTIONS:
Drug: Prednisone — Prednisone 60 mg/m2/day IV over 7 days (-7 a -1) and triple intrathecal therapy (TIT)
Drug: Vincristine — Vincristine (VCR): 1.5 mg/m2 (maximum 2 mg) IV days 1, 8, 15 and 22.
Drug: Daunorubicin — Daunorubicin (DNR): 45 mg/m2 IV days 1, 8, 15 and 22.
Drug: Prednisone — Prednisone (PDN): 60 mg/m2/day, IV or PO, days 1 to 27.
Drug: Ponatinib — Ponatinib 30 mg, PO from day 1 to consolidation
Drug: Mercaptopurine — Mercaptopurine (MP): 50 mg/m2, PO days 1 to 7, 28 to 35 and 56 to 63.
Drug: Methotrexate — MTX: 1,5 g/m2, IV (24 h continuous infusion) days 1, 28 and 56
Drug: VP-16 — VP-16: 100 mg/m2/12 h, IV, days 14 and 42
Drug: ARA-C: — ARA-C: 1000 mg/m2/12 h, IV, days 14-15 and 42-43.
Drug: TIT — TIT (MTX: 12 mg, ARA-C: 30 mg, hydrocortisone: 20 mg), , days 1, 28 and 56.
Drug: Ponatinib — Ponatinib 30 mg/d PO, from day 1 to 15 days before HSCT.
Procedure: Autologous transplantation — Myeloablative conditioning with cyclophosphamide and total body irradiation (TBI) whenever possible and autologous transplantation
Procedure: Allo transplantation — Myeloablative conditioning with cyclophosphamide and total body irradiation (TBI) whenever possible and allo transplantation

SUMMARY:
Evaluate the response (complete hematologic response [CHR], complete cytogenetic response [CCyR], major molecular response [MMR] and complete molecular response [CMR] of the combination of ponatinib with standard chemotherapy (according to PETHEMA ALL Ph08 trial) in young patients with Ph+ (BCR-ABL) ALL.

All patients are treated with:

Pre-phase (maximum 7 days, -7 to -1):

Prednisone 60 mg/m2/day IV over 7 days (-7 a -1) and triple intrathecal therapy (TIT) (Methotrexate [MTX]: 12 mg, ARA-C: 30 mg, hydrocortisone: 20 mg). 2. Induction (day 1 to day 28 or up to hematological recovery) Vincristine (VCR): 1.5 mg/m2 (maximum 2 mg) IV days 1, 8, 15 and 22. Daunorubicin (DNR): 45 mg/m2 IV days 1, 8, 15 and 22. Prednisone (PDN): 60 mg/m2/day, IV or PO, days 1 to 27. Ponatinib 30 mg, PO from day 1 to consolidation. TIT, days 1 and 22. 3. Consolidation (day 1 to day 63) Mercaptopurine (MP): 50 mg/m2, PO days 1 to 7, 28 to 35 and 56 to 63. MTX: 1,5 g/m2, IV (24 h continuous infusion) days 1, 28 and 56. VP-16: 100 mg/m2/12 h, IV, days 14 and 42. ARA-C: 1000 mg/m2/12 h, IV, days 14-15 and 42-43. TIT (MTX: 12 mg, ARA-C: 30 mg, hydrocortisone: 20 mg), , days 1, 28 and 56. Ponatinib 30 mg/d PO, from day 1 to 15 days before HSCT. 4. HSCT (performed ideally within 1 month from the end of consolidation). AlloHSCT preferred over autoHSCT (autoHSCT only indicated if alloHSCT not feasible). Myeloablative conditioning with cyclophosphamide and total body irradiation (TBI) whenever possible. 5. Post HSCT therapy After alloHSCT. Frequent monitoring of MRD (every month). I After autoHSCT: Frequent monitoring of MRD (every month).

DETAILED DESCRIPTION:
Objectives Primary

1. To evaluate the response (complete hematologic response [CHR], complete cytogenetic response [CCyR], major molecular response [MMR] and complete molecular response [CMR] of the combination of ponatinib with standard chemotherapy (according to PETHEMA ALL Ph08 trial) in young patients with Ph+ (BCR-ABL) ALL.
2. To evaluate the event free survival (EFS) of the combination of ponatinib with standard chemotherapy (according to PETHEMA ALL Ph08 trial) in young patients with Ph+ (BCR-ABL) ALL. Secondary

   * To evaluate the rate of patients receiving an allogeneic hematopoietic stem cell transplant (alloHSCT) in first CR
   * To evaluate the frequency of MMR and CMR at the time of alloHSCT
   * To evaluate the transplant-related mortality (TRM)
   * To evaluate the CR duration and overall survival (OS) of the combination of ponatinib with standard chemotherapy (according to PETHEMA ALL Ph08 trial) in young patients with Ph+ (BCR-ABL) ALL.
   * To evaluate the outcome measures (CR duration, OS and EFS) in context of those observed in the PETHEMA ALL Ph08 trial.
   * To observe the type and number of BCR-ABL kinase domain mutations developing during and after the study.
   * To evaluate side effects, adverse events (AE) and serious AE (SAE).

Interventions:

1. Pre-phase (maximum 7 days, -7 to -1):

   Prednisone 60 mg/m2/day IV over 7 days (-7 a -1) and triple intrathecal therapy (TIT) (Methotrexate [MTX]: 12 mg, ARA-C: 30 mg, hydrocortisone: 20 mg).
2. Induction (day 1 to day 28 or up to hematological recovery) Vincristine (VCR): 1.5 mg/m2 (maximum 2 mg) IV days 1, 8, 15 and 22. Daunorubicin (DNR): 45 mg/m2 IV days 1, 8, 15 and 22. Prednisone (PDN): 60 mg/m2/day, IV or PO, days 1 to 27. Ponatinib 30 mg, PO from day 1 to consolidation. TIT, days 1 and 22.
3. Consolidation (day 1 to day 63) Mercaptopurine (MP): 50 mg/m2, PO days 1 to 7, 28 to 35 and 56 to 63. MTX: 1,5 g/m2, IV (24 h continuous infusion) days 1, 28 and 56. VP-16: 100 mg/m2/12 h, IV, days 14 and 42. ARA-C: 1000 mg/m2/12 h, IV, days 14-15 and 42-43. TIT (MTX: 12 mg, ARA-C: 30 mg, hydrocortisone: 20 mg), , days 1, 28 and 56. Ponatinib 30 mg/d PO, from day 1 to 15 days before HSCT.
4. HSCT (performed ideally within 1 month from the end of consolidation). AlloHSCT preferred over autoHSCT (autoHSCT only indicated if alloHSCT not feasible). Myeloablative conditioning with cyclophosphamide and total body irradiation (TBI) whenever possible.
5. Post HSCT therapy After alloHSCT. Frequent monitoring of MRD (every month). If MRD negative: no therapy. If MRD positive, Ponatinib 30 mg/d, po, until 2 yr. after HSCT. The ponatinib dose will be reduced to 15 mg/d in the second year in patients with sustained molecular response. After autoHSCT: Frequent monitoring of MRD (every month). All patients will receive Ponatinib: 30 mg/d, PO, mercaptopurine, (40 mg/m2/d, PO) and methotrexate (15 mg/m2/week, IM), during the first year after HSCT. The ponatinib dose will be reduced to 15 mg/d in the second year in patients with sustained molecular response.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-55 yr.
* De novo Ph+ (BCR-ABL)ALL
* ECOG score ≤2 unless due to ALL
* Absence of significant liver disease, as defined by the following criteria: total serum bilirubin ≤1.5 x upper limit of normal (ULN), unless due to Gilbert's syndrome, alanine aminotransferase (ALT) ≤2.5 × ULN or ≤5 x ULN if leukemic involvement of the liver is present, and aspartate aminotransferase (AST) ≤2.5 × ULN or ≤5 x ULN if leukemic involvement of the liver is present.
* Adequate pancreatic function as defined by serum lipase and amylase ≤1.5 × ULN.
* No history of dyslipidemia, hypertension, thrombotic events or cardiac disease.
* For females of childbearing potential, a negative pregnancy test must be documented prior to randomization. Female and male patients who are fertile must agree to use an effective form of contraception with their sexual partners from randomization through 4 months after the end of treatment.
* informed consent signed, according to national regulation
* Patients aged between 56 and 60 years may be selected who could be included in the study with the authorization of the Coordinating Investigator with the consolidation treatment modified as follows:

Mercaptopurine (MP): 50 mg / m2, PO on days 1 to 7, 28 to 35 and 56 to 63 MTX: 0.75 g / m2, IV (continuous infusion 24 h) on days 1, 28 and 56 ARA-C: 500 mg / m2 / 12 h, IV, days 14-15 and 42-43 TIT (MTX: 12 mg, ARA-C: 30 mg, hydrocortisone: 20 mg), days 1, 28 and 56 Ponatinib 30 mg / d PO, from day 1 to 7 days before HSCT

Exclusion Criteria:

* Lymphoid blast crisis of CML,
* WHO performance status ≤ 50% (Karnofsky) or ≥ 3 (ECOG).
* Active HBV or HCV hepatitis, or AST/ALT ≥ 2.5 x ULN and bilirubin ≥ 1.5 x ULN.
* History of acute pancreatitis within 1 year of study or history of chronic pancreatitis.
* History of alcohol abuse.
* Ongoing or active infections.
* Uncontrolled hypertriglyceridemia (triglycerides >450 mg/dL).
* Clinically significant, uncontrolled or active cardiovascular disease, specifically including, but not restricted to: Any history of myocardial infarction, stroke, or revascularization, Unstable angina or transient ischemic attack within 6 months prior to enrollment Congestive heart failure within 6 months prior to enrollment, or left ventricular ejection fraction (LVEF) less than lower limit of normal per local institutional standards History of clinically significant (as determined by the treating physician) atrial arrhythmia Any history of ventricular arrhythmia Any history of venous thromboembolism including deep venous thrombosis or pulmonary embolism.
* Uncontrolled hypertension (diastolic blood pressure >90 mm Hg; systolic >140 mm Hg). Patients with hypertension should be under treatment on study entry to effect blood pressure control.
* Taking medications that are known to be associated with torsades de pointes.
* Taking any medications or herbal supplements that are known to be strong inhibitors of CYP3A4 within at least 14 days before the first dose of ponatinib.
* Creatinine levels > 2.5mg/dl or glomerular filtration rate (GFR) < 20 ml/min or proteinuria >3.5 g/day.
* Gastrointestinal (GI) function impairment, or a GI disease that may significantly alter the absorption of study drugs.
* Patients who are currently receiving treatment with any of the medications with potential to prolong QT interval (listed in Appendix 4) if the medications cannot be either discontinued or switched to a different medication prior to starting study drug.
* Patients who have received any investigational drug ≤ 4 weeks.
* Patients who have undergone major surgery ≤ 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy.
* Patients who are pregnant or breast feeding and adults of reproductive potential not employing an effective method of birth control (women of childbearing potential must have a negative serum pregnancy test within 48 hrs. prior to administration of Ponatinib). Postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential. Male and female patients must agree to employ an effective barrier method of birth control throughout the study and for up to 4 months following discontinuation of study drugs.
* Patients with a history of another primary malignancy that is currently clinically significant or currently requires active intervention.
* Patients unwilling or unable to comply with the protocol

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2020-08-05 (Actual); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Overall response | 2 years
  To evaluate the response (complete hematologic response [CHR], complete cytogenetic response [CCyR], major molecular response [MMR] and complete molecular response [CMR] of the combination of ponatinib with standard chemotherapy (according to PETHEMA ALL Ph08 trial) in young patients with Ph+ (BCR-ABL) ALL.
Event free survival | 2 years
  To evaluate the event free survival (EFS) of the combination of ponatinib with standard chemotherapy (according to PETHEMA ALL Ph08 trial) in young patients with Ph+ (BCR-ABL) ALL

CONTACTS AND LOCATIONS:
Locations (10):
- Spain (10):
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital Clinic, Barcelona
  - Hospital 12 de Octubre, Madrid
  - Hospital Virgen de la Victoria, Málaga
  - Hospital Clinico Universitario de Salamanca, Salamanca
  - Hospital Marques de Valdecilla, Santander
  - C H Santiago de Compostela, Santiago de Compostela
  - Hospital Virgen del Rocio, Seville
  - Hospital Clinico de Valencia, Valencia
  - Hospital La Fe, Valencia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ribera JM, Garcia-Calduch O, Ribera J, Montesinos P, Cano-Ferri I, Martinez P, Esteve J, Esteban D, Garcia-Fortes M, Alonso N, Gonzalez-Campos J, Bermudez A, Torrent A, Genesca E, Mercadal S, Martinez-Lopez J, Garcia-Sanz R. Ponatinib, chemotherapy, and transplant in adults with Philadelphia chromosome-positive acute lymphoblastic leukemia. Blood Adv. 2022 Sep 27;6(18):5395-5402. doi: 10.1182/bloodadvances.2022007764. PMID 35675590